CLINICAL TRIAL: NCT05297851
Title: Non-interventional Prospective Observational Study of Efficacy and Safety of Cytoflavin in Combination With Reperfusion Compared to Treatment With Other Neuroprotective Drugs Used in Routine Clinical Practice in Patients With Cerebral Infarction
Brief Title: Cytoflavin in Combination With Reperfusion in Stroke Patients
Status: Completed | Type: Observational
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CTF-STRobs-22
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Acute Stroke
Keywords: acute stroke; cerebral infarction; neuroprotection
MeSH Terms: conditions — Stroke; Cerebral Infarction | interventions — cytoflavin; Succinic Acid; Inosine; Niacinamide; Riboflavin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cytoflavin: Patients who underwent reperfusion for acute stroke (intravenous thrombolysis and/or mechanical thrombectomy) and receive intravenous Cytoflavin® at a discretion of the physician, starting this treatment within the first 24 hours from the onset of stroke
  Interventions: Drug: Cytoflavin (succinic acid + inosine + nicotinamide + riboflavin)
- Control: Patients who underwent reperfusion for acute stroke (intravenous thrombolysis and/or mechanical thrombectomy) and do not receive Cytoflavin as part of their routine clinical practice, but may receive any other neuroprotective medications.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Cytoflavin (succinic acid + inosine + nicotinamide + riboflavin) — 10 ml diluted to 100-200 ml of 5-10% dextroseor 0.9% sodium chloride solution. The rate of administration is 3-4 ml / min. The drug is administered in a volume of 10 ml per injection with an interval of 8-12 hours for 10 days. In severe cases of the disease, a single dose is increased to 20 ml.
  Groups: Cytoflavin
Drug: Control — Standard treatment accordind to the routine clinical practice
  Groups: Control

SUMMARY:
Evaluation of the efficacy and safety of Cytoflavin®, solution for intravenous administration, (OOO NTFF POLYSAN, Russia) for 10 days, patients with cerebral infarction who receive reperfusion therapy, with the start of treatment within the first 24 hours from the stroke onset, compared to treament with any other neuroprotective drug which may be used in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent;
2. Men and women 18-85 y.o.;
3. A diagnosis of "cerebral infarction" has been established and treatment with Cytoflavin® has already been prescribed, or other therapy has been prescribed that does not include Cytoflavin®;
4. NIHSS score of at least 5 and less than 24;
5. reperfusion therapy performed on admission;
6. The size of the ischemic focus according to ASPECTS score >=6;
7. Time from stroke onset to admission not exceeeding 6 hours;
8. Start of therapy with Cytoflavin® within 24 hours from the onset of stroke (main group);
9. Patients who are able to follow the procedures of the Observational Study Program and strictly follow the doctor's instructions regarding drug therapy.

Exclusion Criteria:

1. Individual intolerance or known hypersensitivity to succinic acid, inosine, nicotinamide, riboflavin, or auxiliary components of the drug Cytoflavin®;
2. Hemorrhagic stroke;
3. Contraindications for CT scanning;
4. Initial severe disability requiring assistance in everyday life before stroke;
5. previous stroke with a residual neurological deficit;
6. Severe comorbidity with a life expectancy of less than 6 months;
7. Clinical or laboratory signs of an infectious disease on admission (with the exception of strokes that occurred in COVID-19 convalescents after the first 10 days of illness, and patients with asymptomatic SARS-CoV-2 infection detected during routine examination);
8. Pregnancy or lactation

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men and women 18-85 y.o. with acute stroke who receive reperfusion (intravenous thrombolysis and/or mechanical thrombectomy) and continue treatment in the acute stroke unit
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with good functional outcome | 90 days
  Proportion of patients who achieve score 0-2 by modified Rankin scale

CONTACTS AND LOCATIONS:
Overall Officials: Dina R Khasanova, prof., Principal Investigator — Interregional Clinical and Diagnostic Center, Kazan, Russia
Locations (7):
- Russia (7):
  - Northern State Medical University of the Ministry of Health of the Russian Federation, Arkhangelsk
  - Belgorod Regional Clinical Hospital of St. Joasaph, Belgorod
  - Interregional Clinical and Diagnostic Center, Kazan'
  - City Hospital of the Holy Martyr Elizabeth, Saint Petersburg
  - City General Hospital №2, Saint Petersburg
  - City Mariinsky Hospital, Saint Petersburg
  - SPb GBUZ "City Hospital №26", Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided